CLINICAL TRIAL: NCT00760071
Title: Evaluation of Morphological and Functional Magnetic Resonance Imaging (MRI) for Early Diagnosis of Lung Changes in Children (0-6 Years) With Cystic Fibrosis (CF)
Brief Title: Magnetic Resonance Imaging (MRI) for Early Diagnosis of Cystic Fibrosis (CF)
Status: Completed | Type: Observational
Sponsor: German Cancer Research Center (Other)
Collaborators: Mukoviszidose Institut gGmbH (Other); Heidelberg University (Other)
Responsible Party: German Cancer Research Center, Helmholz society
Other Study IDs: 387/2005
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Last update posted 2010-04-15 (Estimated); Status verified 2010-04

CONDITIONS: Cystic Fibrosis; Lung Disease
Keywords: cystic fibrosis,; lung disease,; MRI,; morphology,; function; morphological MRI; functional MRI; correlation to clinical data
MeSH Terms: conditions — Cystic Fibrosis; Lung Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1CF-patients<6: Patients with diagnoses of cystic fibrosis from birth to the age of 6 years
- 2 controls: age matched controls

SUMMARY:
In patients with Cystic Fibrosis (CF) the clinical course of lung disease is crucial for individual prognosis and life expectancy.

Imaging modalities are important in the assessment of follow up of structural lung changes and monitoring of pulmonary complications in CF. Although high resolution computed tomography (HRCT) is the accepted gold standard for evaluation of morphological lung changes in CF, chest-X-ray is widely used as standard imaging procedure for assessment and follow up in these young patients due to less radiation exposure.

Magnetic resonance imaging (MRI) has not been used for lung imaging in CF so far. Studies from the 80's and early 90's were not able to show any impact for the use of MRI in CF. Due to recent technical developments MRI of the lung became possible.

Our study group was able to show that MRI is a competitive imaging modality for evaluating changes of the CF-lung in comparison to the gold standard (HRCT).

So far only patients from the age of 6-7 years were examined. According to recent studies CF is a disease which starts in utero. Therefore it can lead to extensive pulmonary changes even in infants and young children. In this age group lung function testing is difficult and not broadly available. An early optimized therapy is crucial for the long term course and outcome of the pulmonary disease.

The aim of this study is to evaluate morphological and functional MRI for early diagnosis of lung changes in children (0-6 years) with CF.

DETAILED DESCRIPTION:
Month 1-2: Protocol adaptation for infants and small children Month 3-14: Patient examinations (20 Patients with sedation) Month 15-18: Data evaluation

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the parents or a legal guardian
* Sedation as necessary
* Conventional clinical indicated diagnostic procedures (lung function test, chest-X-ray, CT)

Exclusion Criteria:

* Study exclusion in case of contra indications for MRI:

  * Patients with cardiac pace maker, metallic implants (e.g. cerebral vessel clips) as well as other conditions that prohibit the exposition of a patient to a strong magnetic field.
  * No informed consent
  * Dyspnea, which disables the patient to follow breathing instructions during the study.

Ages: 1 Day to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Diagnosed CF-patients (male/female), age 0-6 years
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-10 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Puderbach, MD, Principal Investigator — German Cancer Research Center
Locations (1):
- German Cancer Research Center, Heidelberg, Germany

REFERENCES:
- [Derived] Wielputz MO, Stahl M, Triphan SMF, Wucherpfennig L, Leutz-Schmidt P, Gestewitz S, Steinke E, Graeber SY, Kauczor HU, Eichinger M, Puderbach MU, Alrajab A, Schenk JP, Sommerburg O, Mall MA. Longitudinal Magnetic Resonance Imaging of Changes in Lung Morphology and Perfusion in Children with Cystic Fibrosis from Infancy through Adolescence. Ann Am Thorac Soc. 2025 Jan;22(1):93-103. doi: 10.1513/AnnalsATS.202404-396OC. PMID 39255452
- [Derived] Sommerburg O, Wielputz MO, Trame JP, Wuennemann F, Opdazaite E, Stahl M, Puderbach MU, Kopp-Schneider A, Fritzsching E, Kauczor HU, Baumann I, Mall MA, Eichinger M. Magnetic Resonance Imaging Detects Chronic Rhinosinusitis in Infants and Preschool Children with Cystic Fibrosis. Ann Am Thorac Soc. 2020 Jun;17(6):714-723. doi: 10.1513/AnnalsATS.201910-777OC. PMID 32142375
- [Derived] Wielputz MO, Puderbach M, Kopp-Schneider A, Stahl M, Fritzsching E, Sommerburg O, Ley S, Sumkauskaite M, Biederer J, Kauczor HU, Eichinger M, Mall MA. Magnetic resonance imaging detects changes in structure and perfusion, and response to therapy in early cystic fibrosis lung disease. Am J Respir Crit Care Med. 2014 Apr 15;189(8):956-65. doi: 10.1164/rccm.201309-1659OC. PMID 24564281
- See also: German Cystic Fibrosis Foundation — http://muko.info/